CLINICAL TRIAL: NCT01417156
Title: A Phase II Open Label, Follow up Study to Investigate the Long Term Tolerability and Safety of Oral BIBF 1120 on Top of Pirfenidone in Japanese Patients With Idiopathic Pulmonary Fibrosis
Brief Title: Safety and PK Study of BIBF 1120 in Japanese Patients With IPF: Follow up Study From 1199.31(NCT01136174)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1199.40
Record Dates: First submitted 2011-08-15; First posted 2011-08-16 (Estimated); Results first posted 2017-03-06 (Actual); Last update posted 2017-03-06 (Actual); Status verified 2017-01

CONDITIONS: Pulmonary Fibrosis
MeSH Terms: conditions — Pulmonary Fibrosis | interventions — nintedanib

ARMS (1):
- All patients (Experimental)
  Interventions: Drug: Nintedanib; Drug: Pirfenidoneone

INTERVENTIONS:
Drug: Nintedanib — 150 mg bid
Drug: Pirfenidoneone — Existing treatment

SUMMARY:
Primary objective of this study is to investigate the long-term tolerability and safety profile of BIBF 1120 on top of pirfenidone treatment in patients with Idiopathic Pulmonary Fibrosis who have completed a prior clinical trial of BIBF 1120 (1199.31).

Secondary objectives are to assess effects on some efficacy criteria during long term treatment with BIBF 1120 on top of pirfenidone.

ELIGIBILITY:
Inclusion criteria:

1. Written informed consent consistent with Good Clinical Practice (GCP) signed prior to entry into the study
2. Completion of 1199.31 study and still under treatment with pirfenidone at a stable dose

Exclusion criteria:

1. Any disease that may interfere with testing procedures or in judgement of investigator may interfere with trial participation or may put the patient at risk when participating in this trial. Reconsider carefully all exclusion criteria of trial 1199.31. However, patients may qualify for participation even though they meet the exclusion criteria (for 1199.31), if the investigators benefit-risk assessment remains favorable.
2. Any other investigational therapy received within 8 weeks before visit 1.
3. For female: Pregnant women or women who are breast feeding or of child bearing potential not using a highly effective method of birth control for both at least 4 weeks prior to enrolment and 10 weeks after last study drug intake.

   For male: Sexually active males not committing to using condoms both during the course of the study and ten weeks after last study drug intake (except if their partner is not of childbearing potential).
4. Known or suspected active alcohol or drug abuse.
5. Patients who require full-dose therapeutic anticoagulation (e.g. vitamin K antagonists, heparin), except low dose heparin and/or heparin flash as needed for maintenance of an indwelling intravenous device. As an example, prophylactic use of heparin, e.g. enoxaparin 2000 International unit (I.U.) subcutaneously (s.c.) per day, should be allowed.
6. Patients who require full-dose antiplatelet (e.g. acetyl salicylic acid, clopidogrel) therapy. As an example, chronic low-dose acetyl salicylic acid, below or equal to 100 mg per day, should be allowed.
7. Patient not compliant in previous trial, with trial medication or trial visits.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (4):
- Japan (4):
  - Boehringer Ingelheim Investigational Site, Himeji, Hyogo
  - Boehringer Ingelheim Investigational Site, Sakai, Osaka
  - Boehringer Ingelheim Investigational Site, Seto, Aichi
  - Boehringer Ingelheim Investigational Site, Yokohama, Kanagawa

RESULTS

PARTICIPANT FLOW:
Groups:
- Nintedanib: Patients were treated orally with 150 milligram (mg) Nintedanib (BIBF 1120) twice daily (b.i.d.) on top of pre-existing Pirfenidone treatment with the opportunity to reduce the dose to 100 mg bid to manage adverse events.
Period: Overall Study
Arm/Group | Nintedanib
Started | 20
Completed | 6
Not Completed | 14
Not completed — Adverse Event | 12
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Population: Treated set (TS): This analysis set included all patients who were given study medication and were documented to have taken at least one dose of the trial medication.
Arm/Group | Nintedanib
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.8 (9.5)
Gender [Count of Participants; unit: Participants]
  Female | 6
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Overall Adverse Events
Description: Incidence (Number of patients) of Adverse events (AEs) over the course of treatment period including serious adverse events (SAEs), AEs leading to discontinuation of study medication, and fatal AEs.
Time Frame: First drug administration until end of treatment, up to 5 years
Population: Treated set (TS)
Measure: Number; unit: participants
Arm/Group | Nintedanib
Number analyzed (Participants) | 20
participants
  AEs leading to discontinuation of trial drug | 12
  Fatal | 8
  Severe AEs | 11

2. Secondary Outcome: Annual Rate of Decline in Forced Vital Capacity (FVC).
Description: The adjusted annual rate of decline in Forced Vital Capacity (FVC). The means presents actually the adjusted rate based on a random coefficient regression with fixed effects for gender, age, height and random effect of patient specific intercept and time. Within-patient errors are modelled by an Unstructured variance-covariance matrix. Inter-individual variability is modelled by a Variance-Components variance-covariance matrix.
  The result for Annual rate of decline (ROD) in FVC should be interpreted with caution and along with descriptive statistics, because inferences used for this analysis might not be valid as suggested by skewed distribution of the data.
Time Frame: Baseline and every 8 weeks after drug administration until end of treatment, up to 5 years
Population: TS-OC Observed Case (OC): This method was used for the replacement of missing values.
Measure: Least Squares Mean (Standard Error); unit: (mililitre (mL)/year)
Arm/Group | Nintedanib
Number analyzed (Participants) | 20
(mililitre (mL)/year) | -233.3 (72.59)

3. Secondary Outcome: Annual Rate of Decline in Haemoglobin (Hb) Corrected Diffusing Capacity of the Lung for Carbon Monoxide (DLCO)
Description: Adjusted annual rate of decline in Hb corrected DLCO. The means presents actually adjusted rate based on random coefficient regression with fixed effects for gender, age, height & random effect of patient specific intercept & time. Within-patient errors are modelled by Unstructured variance-covariance matrix.Inter-individual variability is modelled by a variance-Components variance-covariance matrix.
  mmHg: millimeters of mercury
Time Frame: Baseline & every 8 weeks after drug administration until end of treatment, up to 5 years
Population: OC-TS
Measure: Mean (Standard Error); unit: mL/Minute(min)/mmHg per year
Arm/Group | Nintedanib
Number analyzed (Participants) | 20
mL/Minute(min)/mmHg per year | -1.3 (0.26)

4. Secondary Outcome: Acute Exacerbations of IPF: Risk (Incidence Rate) of Acute Exacerbations of IPF.
Description: The risk (incidence rate calculated as number of patients with at least 1 exacerbation, divided by the total time at risk ×100) of acute exacerbation of IPF.
Time Frame: First drug administration until end of treatment, up to 5 years
Population: TS
Measure: Number (95% Confidence Interval); unit: patients per 100 patient-year
Arm/Group | Nintedanib
Number analyzed (Participants) | 20
patients per 100 patient-year | 19.2 [8.29 to 37.82]

5. Secondary Outcome: Percentage of Patient With First Occurrence of Acute Exacerbations of Idiopathic Pulmonary Fibrosis (IPF) Until Week 234.
Description: The percentage of patient having first acute exacerbation of Idiopathic Pulmonary Fibrosis (IPF) based on investigator reported adverse events until week 234.
Time Frame: Week 234
Population: TS
Measure: Number; unit: percentage of participants
Arm/Group | Nintedanib
Number analyzed (Participants) | 20
percentage of participants
  Failure (Week 234) | 40.0
  Censored (Week 234) | 60.0

ADVERSE EVENTS:
Time Frame: First drug administration until end of treatment, up to 5 years
Arm/Group | Nintedanib
Serious Adverse Events (participants affected / at risk) | 16/20
Other Adverse Events (participants affected / at risk) | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib (N=20)
Acute myocardial infarction (Cardiac disorders) | 1
Right ventricular failure (Cardiac disorders) | 1
Anal fistula (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Pyrexia (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 2
Appendicitis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Respiratory tract infection (Infections and infestations) | 2
Tuberculosis (Infections and infestations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 2
Tendonitis (Musculoskeletal and connective tissue disorders) | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 13
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2
Deep vein thrombosis (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib (N=20)
Anaemia (Blood and lymphatic system disorders) | 2
Abdominal discomfort (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 4
Abdominal pain upper (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 8
Dental caries (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 13
Gastritis (Gastrointestinal disorders) | 2
Haemorrhoids (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 12
Vomiting (Gastrointestinal disorders) | 5
Chest pain (General disorders) | 2
Oedema peripheral (General disorders) | 2
Pyrexia (General disorders) | 3
Bronchitis (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 7
Oral candidiasis (Infections and infestations) | 3
Pharyngitis (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 2
Hepatic enzyme increased (Investigations) | 3
Weight decreased (Investigations) | 5
Decreased appetite (Metabolism and nutrition disorders) | 7
Hyperkalaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3
Dysgeusia (Nervous system disorders) | 3
Headache (Nervous system disorders) | 2
Insomnia (Psychiatric disorders) | 4
Haematuria (Renal and urinary disorders) | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 2
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2
Eczema (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 6

LIMITATIONS AND CAVEATS:
Annual ROD in FVC results to be interpreted with caution & along with descriptive statistics as inferences used might not be valid as suggested by skewed distribution of data thus Absolute Change from baseline in FVC over time has been defined.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.